CLINICAL TRIAL: NCT04119583
Title: Efficacy of an U-shape Automatic Electric Toothbrush in Plaque Removal: a Crossover Randomized Study
Brief Title: Efficacy of an U-shape Automatic Electric Toothbrush in Plaque Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Lorenzo Franchi, Associate Professor in Dentistry, University of Florence
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IUFET1
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Dental Plaque; Toothbrushing
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- U-shape Automatic Electric Toothbrush (Experimental)
  Interventions: Device: U-shape Automatic Electric Toothbrush
- Usual home toothbrushing procedure (Active Comparator)
  Interventions: Other: Usual home toothbrushing procedure
- No toothbrushing (No Intervention)
- Conventional Electric Toothbrush (Active Comparator)
  Interventions: Other: Conventional Electric Toothbrush

INTERVENTIONS:
Device: U-shape Automatic Electric Toothbrush — The U-shape Automatic Electric Toothbrush will be applied for 30-45 seconds on the teeth of both arches without the use of toothpaste.
  Arms: U-shape Automatic Electric Toothbrush
Other: Usual home toothbrushing procedure — Usual home toothbrushing procedure either with manual or electric toothbrush without the use of toothpaste.
  Arms: Usual home toothbrushing procedure
Other: Conventional Electric Toothbrush — The Conventional Electric Toothbrush will be applied for 2 minutes on the teeth of both arches without the use of toothpaste.
  Arms: Conventional Electric Toothbrush

SUMMARY:
Over time, many different types of manual and electric toothbrushes have been produced. A systematic review has shown that some electric toothbrushes are more effective at removing bacterial plaque than manual toothbrushes. A new U-shaped electric toothbrush with silicone bristles has recently been produced that has a fully automatic and simultaneous action on both arches. However, its efficacy in removing bacterial plaque is not clear at the moment, as no randomized study has been published on this type of toothbrush.

The aim of this study is to compare the efficacy in terms of bacterial plaque removal in a single use of a new automatic U-shaped electric toothbrush, compared with the usual home toothbrushing procedure, a conventional electric toothbrush, and negative control (no toothbrushing) in a group of volunteer students of the School of Dentistry of the University of Florence, Italy.

Primary endpoint will be the difference in "full mouth plaque score" between before and after brushing. Secondary endpoints will be feeling of "clean mouth" evaluated on a VAS (Visual Analogue Scale) scale from 0 to 10 where 0 indicates no feeling of clean mouth and 10 maximum feeling of clean mouth.

This study will be a monocentric, randomized, controlled, superiority, cross-over study, with blind examiner and 4 therapies (U-shaped electric toothbrush, usual home toothbrushing procedure, conventional electric toothbrush, no toothbrushing), carried out in a single session with an interval of one week between the 4 therapies.

Study population will be students of the School of Dentistry who are healthy volunteers. Number of patients to be enrolled: 22. Inclusion criteria: age between 18 and 30 years; no fixed orthodontic appliance; presence of at least 20 teeth; Full mouth plaque score (FMPS) above 40%.

Exclusion criteria: subjects with manual disabilities to perform normal oral hygiene maneuvers; subjects allergic to silicone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years;
* no fixed orthodontic equipment;
* presence of at least 20 teeth;
* Full mouth plaque score (FMPS) above 40%.

Exclusion Criteria:

* Subjects with manual disabilities to perform normal oral hygiene maneuvers;
* Subjects allergic to silicone

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Full mouth plaque score | Difference between pre- and post-brushing (time frame 10-15 minutes)
  Percentage of sites that presents with plaque on the total of the sites examined (6 sites per tooth).

SECONDARY OUTCOMES:
Feeling of "clean mouth" | Post-brushing (time frame 1-2 minutes)
  Visual analogue scale from 0 to 10 where 0 indicates no feeling of clean mouth and 10 maximum feeling of clean mouth

CONTACTS AND LOCATIONS:
Locations (1):
- SOD Odontostomatologia, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided